CLINICAL TRIAL: NCT07271849
Title: Effects of Different Administration Timings of Nalbuphine on Hemodynamics and Postoperative Analgesia in Elderly Patients Undergoing Total Knee Arthroplasty
Brief Title: Nalbuphine Timing Effects on Hemodynamics and Analgesia in Elderly Patients
Acronym: TKA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Liang Guo, The First Affiliated Hospital of Shandong First Medical University (Shandong Provincial Qianfoshan Hospital), Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: YXLL-KY-2025(207)
Record Dates: First submitted 2025-11-17; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain, Acute; Hemodynamics; Total Knee Arthroplasty (TKA)
Keywords: Total Knee Arthroplasty (TKA); Postoperative Pain; Nalbuphine; Hemodynamics
MeSH Terms: conditions — Pain, Postoperative | interventions — Nalbuphine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group N0 (Experimental): Anesthesia Induction: Dexamethasone (10 mg), midazolam (0.01-0.05 mg/kg), sufentanil (0.2-0.4 μg/kg), etomidate (0.15-0.3 mg/kg), and atracurium (0.3-0.6 mg/kg) were administered intravenously. After complete neuromuscular blockade was achieved, a laryngeal mask airway was inserted (size selected according to body weight).Intravenous nalbuphine (0.2 mg/kg) was administered during anesthesia induction. Anesthesia was maintained by continuous intravenous infusion of propofol (4-12 mg/kg/h) and remifentanil (0.15-0.3 μg/kg/min)
  Interventions: Drug: Nalbuphine Hydrochloride injection was administered during anesthesia induction.
- Group N1 (Experimental): Anesthesia Induction: Dexamethasone (10 mg), midazolam (0.01-0.05 mg/kg), sufentanil (0.2-0.4 μg/kg), etomidate (0.15-0.3 mg/kg), and atracurium (0.3-0.6 mg/kg) were administered intravenously. After complete neuromuscular blockade was achieved, a laryngeal mask airway was inserted (size selected according to body weight).Intravenous nalbuphine (0.2 mg/kg) was administered after cement implantation. Anesthesia was maintained by continuous intravenous infusion of propofol (4-12 mg/kg/h) and remifentanil (0.15-0.3 μg/kg/min).
  Interventions: Drug: Nalbuphine Hydrochloride injection was administered after cement implantation.
- Control Group (Group C) (Active Comparator): Anesthesia Induction: Dexamethasone (10 mg), midazolam (0.01-0.05 mg/kg), sufentanil (0.2-0.4 μg/kg), etomidate (0.15-0.3 mg/kg), and atracurium (0.3-0.6 mg/kg) were administered intravenously. After complete neuromuscular blockade was achieved, a laryngeal mask airway was inserted Conventional induction and anesthesia was maintained by continuous intravenous infusion of propofol (4-12 mg/kg/h) and remifentanil (0.15-0.3 μg/kg/min) were performed, with no intravenous nalbuphine administered for analgesia.
  Interventions: Other: Standard general anesthesia regimen ( nalbuphine was not administered throughout the entire anesthesia process.)

INTERVENTIONS:
Drug: Nalbuphine Hydrochloride injection was administered during anesthesia induction. — A single intravenous injection of Nalbuphine Hydrochloride Injection (dose specified, e.g., 0.2 mg/kg) was administered to the patient during general anesthesia induction. Neither the control group nor intervention group N1 received the drug during this stage.The remainder of the anesthesia protocol was consistent across all three groups.
  Other Names: Nalbuphine
  Arms: Group N0
Drug: Nalbuphine Hydrochloride injection was administered after cement implantation. — After intraoperative prosthesis placement, a single intravenous injection of nalbuphine hydrochloride injection (0.2 mg/kg), identical to that in Intervention Group N0) was administered. Neither the control group nor Intervention Group N0 received medication at this timing. All other anesthesia management procedures were standardized.
  Other Names: Nalbuphine
  Arms: Group N1
Other: Standard general anesthesia regimen ( nalbuphine was not administered throughout the entire anesthesia process.) — Conventional induction and anesthesia was maintained were performed, with no intravenous nalbuphine administered for analgesia.
  Arms: Control Group (Group C)

SUMMARY:
In total knee arthroplasty (TKA), the use of a tourniquet and controlled hypotension is common. However, ischemia-reperfusion injury induced by the tourniquet and inappropriate controlled hypotension can lead to cardiac and cerebral damage in patients. Consequently, maintaining hemodynamic stability, ensuring adequate cerebral perfusion, and achieving controlled blood pressure during the perioperative period are critical factors influencing patient outcomes. Postoperatively, patients typically experience moderate to severe pain. Severe postoperative pain can result in prolonged hospital stays, increased readmission rates, elevated opioid consumption, and associated nausea and vomiting. Therefore, exploring effective multimodal postoperative pain management strategies is essential. Nalbuphine, an opioid analgesic acting as a full kappa-receptor agonist and a partial mu-receptor antagonist, is considered to provide analgesic efficacy equivalent to morphine while potentially offering advantages in maintaining hemodynamic stability. This study aims to investigate the effects of administering equivalent doses of nalbuphine at different perioperative time points on analgesia and hemodynamics in elderly patients undergoing knee arthroplasty.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a widely performed routine surgical procedure for treating end-stage osteoarthritis (OA) or rheumatoid arthritis, aiming to alleviate pain and improve the quality of life for participants . However, participants undergoing TKA frequently experience moderate to severe postoperative pain during the perioperative period, with some even suffering from extremely severe pain . Intense postoperative pain can lead to prolonged hospital stays, increased readmission rates, elevated opioid consumption, and associated complications such as nausea and vomiting. These factors diminish participant satisfaction and escalate healthcare costs . Consequently, effective postoperative pain management is crucial for promoting early recovery and improving participant outcomes.

During TKA, periarticular tissue dissection and osteotomy cause bleeding and traumatic inflammation. Techniques such as tourniquet application and controlled hypotension are commonly employed. However, tourniquet-induced ischemia-reperfusion injury and inappropriate controlled hypotension can result in cardiac and cerebral injury for participants. Therefore, maintaining hemodynamic stability, ensuring adequate cerebral perfusion, and achieving controlled blood pressure throughout the perioperative period are critical factors for participant prognosis .

Opioids remain the conventional medication for perioperative pain relief. While effective for analgesia, they are associated with adverse effects such as respiratory depression, postoperative nausea and vomiting (PONV), and pruritus. Nalbuphine, an opioid acting as a full κ-receptor agonist and partial μ-receptor antagonist, is considered to provide analgesic efficacy equivalent to morphine and is widely used for managing moderate to severe postoperative pain . Studies indicate that nalbuphine offers superior hemodynamic stability and analgesic effects compared to morphine across various surgical procedures. It not only alleviates postoperative pain but also demonstrates a lower incidence of PONV. Its analgesic and sedative properties are also considered safe for use in pediatric populations . Nevertheless, conclusive evidence regarding the analgesic and hemodynamic effects of nalbuphine in elderly participants undergoing knee arthroplasty during the perioperative period remains lacking.

Therefore, this study aims to investigate the impact of administering equivalent doses of nalbuphine at different perioperative time points on analgesia and hemodynamics in elderly participants undergoing total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* All study participants voluntarily enrolled in the trial and provided written informed consent after being fully informed of the trial's purpose and significance
* Participants underwent unilateral total knee arthroplasty under general anesthesia
* Elderly participants (age ≥ 65 years), regardless of gender
* Body mass index (BMI) ranging from 18 kg/m² to 30 kg/m²
* Absence of psychiatric disorders, normal consciousness, and ability to communicate effectively
* American Society of Anesthesiologists (ASA) physical status classification I-III;
* No contraindications to the study medications

Exclusion Criteria:

* Study participants with uncontrolled or untreated hypertension (resting systolic/diastolic blood pressure >180/100 mmHg)
* Individuals with severe respiratory diseases
* Subjects with abnormal liver or renal function (ALT and/or AST >2.5 times the upper limit of normal, total bilirubin >1.5 times the upper limit of normal, serum creatinine >1.5 times the upper limit of normal)
* Individuals with a history of drug abuse, illicit drug use, or alcohol abuse, where alcohol abuse is defined as an average daily alcohol intake exceeding 2 units (1 unit = 360 mL of beer, 45 mL of 40% alcohol by volume spirits, or 150 mL of wine)

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) scores of participants at 30 minutes postoperatively. | at 30 minutes postoperatively
  VAS (Visual Analogue Scale) is a tool used to quantify subjective pain intensity via a visual linear scale. Its core design involves a 10 cm straight line, with the left end marked "no pain" (0 points) and the right end "severe pain" (10 points). Patients mark a position on the line based on their perceived pain, and clinicians convert this to a 0-10 pain score by measuring the distance (in millimeters) from the marked point to the left end.

SECONDARY OUTCOMES:
Hemodynamic parameters at various perioperative time points， Parameters include blood pressure, mean arterial pressure (MAP) | T0 (during anesthesia induction), T1 (5 minutes after induction ), T2 (before cement placement), T3 (5 minutes after cement placement), T4 (15minutes post-anesthesia ), T5 (15 minutes in the Post-Anesthesia Care Unit, PACU), and T6 (30 minutes in PACU).
  Blood pressure is the lateral pressure exerted by blood on the walls of blood vessels during circulation, consisting of systolic pressure (when the heart contracts) and diastolic pressure (when the heart relaxes).
Hemodynamic parameters at various perioperative time points，heart rate (HR). | T0 (during anesthesia induction), T1 (5 minutes after induction ), T2 (before cement placement), T3 (5 minutes after cement placement), T4 (15minutes post-anesthesia ), T5 (15 minutes in the Post-Anesthesia Care Unit, PACU), and T6 (30 minutes in PACU).
  Heart rate refers to the number of heartbeats per minute
Postoperative pain assessment using the Visual Analog Scale (VAS) | after extubation, and at 30 minutes, 2 hours, 4 hours, 8 hours, 12 hours, and 24 hours postoperatively.
  VAS (Visual Analogue Scale) is a tool used to quantify subjective pain intensity via a visual linear scale. Its core design involves a 10 cm straight line, with the left end marked "no pain" (0 points) and the right end "severe pain" (10 points). Patients mark a position on the line based on their perceived pain, and clinicians convert this to a 0-10 pain score by measuring the distance (in millimeters) from the marked point to the left end.
Requirement for rescue analgesic medication within 24 hours postoperatively | within 24 hours postoperatively:
  The cumulative Opioids consumption such as demerol,sufentanil,morphine
the number of participants requiring rescue analgesia | within 24 hours postoperatively
  The number of patients who required additional analgesics such as opioids(demerol,sufentanil,morphine)or non-steroid anti-inflammatory drugs(acetaminophen,diclofenac).
Incidence of adverse reactions within 24 hours postoperatively | within 24 hours postoperatively
  (Postoperative nausea and vomiting)Nausea is defined as subjective,unpleasant sensation associated with awareness of the urge to vomit. Retching is defined as the laboured, spastic, rhythmic contraction of the respiratory muscles without expulsion of the gastric contents.Vomiting is defined as the forceful expulsion of gastric contents from the mouth.The adverse central nervous system (CNS) events(such as nightmares, hallucinations, dizziness, itchy skin) were recorded (yes/no).
The types and dosages of vasoactive drugs administered to patients during the perioperative period were recorded | at 30 minutes postoperatively
  If non-invasive blood pressure exceeded the patient's baseline value by 10%, urapidil hydrochloride injection was administered; if it was lower than the baseline by 10%, norepinephrine was administered. The types and dosages of vasoactive drugs used in each group were promptly documented.
The surgical duration time | Immediately after surgery
  The surgical duration was defined as the period from the surgeon's initial skin incision to the completion of skin closure.
The time of laryngeal mask airway (LMA) removal were recorded. | 10-15 minutes after the conclusion of the surgery.
  LMA removal was performed when the patient regained consciousness and maintained SpO₂ above 90% while breathing room air spontaneously for 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Guo Liang, Ph.D, Principal Investigator — Qianfoshan Hospital
Locations (1):
- Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University,, Jinan, Shandong, China